CLINICAL TRIAL: NCT02010060
Title: The Intervention Composed of Aerobic Training and Non-Exercise Physical Activity (I-CAN)
Brief Title: Aerobic Training and Non-Exercise Physical Activity
Acronym: I-CAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Damon Swift, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13SDG17140091
Record Dates: First submitted 2013-12-05; First posted 2013-12-12 (Estimated); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Central Obesity; Obesity
Keywords: Exercise training; Non-exercise physical activity; pedometers
MeSH Terms: conditions — Obesity, Abdominal; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): The goal of this group is to maintain their current lifestyle habits during the intervention. participants are asked to make no conscious changes to their physical activity or dietary habits.
- Aerobic Exercise Training (Experimental): The Aerobic training group will participate in 6 months of aerobic training and asked to make no conscious alterations in their physical activity outside of exercise session, or dietary habits
  Interventions: Behavioral: Aerobic Exercise Training
- Aerobic Exercise+ Physical Activity (Experimental): The goal of this group is to perform 6 months of aerobic exercise and increase the amount of physical activity outside of their training sessions. They will be asked to make no conscious changes to their dietary habits
  Interventions: Behavioral: Aerobic Exercise+ Physical Activity

INTERVENTIONS:
Behavioral: Aerobic Exercise Training — Individuals randomized to the aerobic exercise training group will participate in 6 months of supervised exercise training. Exercise dose (expressed in kilocalories per kg per week [KKW]) during aerobic training will be 8KKW in week 1, 10KKW in week 2 and 12 KKW in week 3. the exercise dose of 12KKW will be maintained throughout the intervention. Pedometers will be worn by participant in blind-mode throughout the intervention, and removed during exercise training sessions. Participants will enter information about whether they wore their pedometer on the study website. Aerobic exercise group participants will be told to make no conscious alterations to their physical activity or dietary habits
  Arms: Aerobic Exercise Training
Behavioral: Aerobic Exercise+ Physical Activity — The Aerobic Exercise+ Physical Activity Group will participate in the same supervised exercise training intervention as the Aerobic Exercise Group, but will also increase the amount of non-exercise physical activity in their daily lives. After week 6 of intervention, participants will incrementally increase Non-Ex PA until they reach an average of 3,000 steps/day above baseline. Non-Ex PA will be increased with moderate physical activity consistent with daily living (i.e. leisurely walking in the evening, walking the dog etc.). Participants will also periodically have life-style counseling sessions with instructors with expertise in behavioral change support to their dietary habits
  Arms: Aerobic Exercise+ Physical Activity

SUMMARY:
This study will determine the health benefits of combining exercise training and increasing the amount of physical activity in daily life on the fat around the abdomen, weight, fitness and sensitivity to insulin. Volunteers will participate in one of three groups for 6 months: 1) a control group, 2) exercise training only, or 3) exercise training and increasing physical activity outside of training. The exercise training will follow the public health recommendations for exercise (150 minutes/week of moderate exercise). The group increasing physical activity along with exercise training will be asked to increase physical activity in their daily life (up to 3,000 step/day above their current levels through the use of step counters), and meetings focused on behavior modification. The investigators hypothesize that combining aerobic training and additional physical activity after training will have the most profound reduction on waist circumference and body composition.

DETAILED DESCRIPTION:
The Intervention Composed of Aerobic Training and Non-Exercise Physical Activity (I-CAN) study will investigate the effects of aerobic exercise training and increasing the amount of physical activity outside of training (Non-EX PA) on waist circumference, weight, and other cardiovascular disease risk factors in a prospective pilot trial. The investigators will randomize sedentary (<6,500 steps per day) obese adults with at least one additional cardiovascular risk factor (N= 45) to a: (1) structured aerobic exercise program with no intervention on Non-Ex PA (AERO group, N=15); (2) structured aerobic exercise program with the additional goal of increasing Non-EX PA (AERO-PA group, N=15), or (3) a non-exercise control group (CON, N=15) for 6 months. Exercise groups will participate in the same aerobic training program (50 to 75% VO2 max), designed to be consistent with public health recommendations of 150 minutes per week of moderate physical activity. Non-Ex PA in the AERO group will be tracked throughout the entire 6 month intervention with pedometers capable of counting steps, but not displaying them to the participant (blind mode capable). The AERO-PA group will progressively increase Non-Ex PA throughout intervention using pedometers (a progressive increase of 1,000 to 3,000 steps per day above baseline levels). The AERO-PA group will also participate in lifestyle counseling grounded in the principles of the behavioral change theories to determine/reinforce strategies to increase Non-Ex PA. The primary outcome measure will be change in waist circumference following the intervention. The results of this pilot study will be used to determine the efficacy/feasibility of the intervention, and power a larger trial as an R01 application.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 65 years
* Body mass index: 30-40
* Sedentary status
* One additional risk factor for cardiovascular disease
* High waist circumference

Exclusion Criteria:

* Previous heart attack or stroke
* Type 1 or type 2 diabetes
* Resting systolic blood pressure >180 mmHg
* Resting diastolic blood pressure>100 mmHg
* Plans to be away from the Pitt County area more than 4 weeks in the next 6 months
* Currently pregnant or plans to become pregnant
* Not full-filling requirements during the screening process
* Currently using weight loss medications
* Gastric banding surgery

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damon L Swift, Ph.D., Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swift DL, Dover SE, Nevels TR, Solar CA, Brophy PM, Hall TR, Houmard JA, Lutes LD. The intervention composed of aerobic training and non-exercise physical activity (I-CAN) study: Rationale, design and methods. Contemp Clin Trials. 2015 Nov;45(Pt B):435-442. doi: 10.1016/j.cct.2015.11.005. Epub 2015 Nov 2. PMID 26542389
- [Derived] Swift DL, Nevels TR, Solar CA, Brophy PM, McGee JE, Brewer SB, Clark A, Houmard JA, Lutes LD. The Effect of Aerobic Training and Increasing Nonexercise Physical Activity on Cardiometabolic Risk Factors. Med Sci Sports Exerc. 2021 Oct 1;53(10):2152-2163. doi: 10.1249/MSS.0000000000002675. PMID 33867498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the local Greenville, NC area. Participants were recruited through flyers, the local newspaper, and email list in the Greenville area.
Pre-assignment Details: Participant could be excluded from enrollment prior to randomization if they do not meet the criteria for enrollment, failure to comply with the requirements of the study pre-enrollment period (e.g. do not schedule study visit) or medical issues are discovered during the screening process that would make them ineligible for enrollment.
Groups:
- Control (CON): The goal of this group is to maintain their current lifestyle habits during the intervention. participants are asked to make no conscious changes to their physical activity or dietary habits.
- Aerobic Exercise Training (AERO): The Aerobic training group will participate in 6 months of aerobic training and asked to make no conscious alterations in their physical activity outside of exercise session, or dietary habits
  Aerobic Exercise Training: Individuals randomized to the aerobic exercise training group will participate in 6 months of supervised exercise training. Exercise dose (expressed in kilocalories per kg per week [KKW]) during aerobic training will be 8KKW in week 1, 10KKW in week 2 and 12 KKW in week 3. the exercise dose of 12KKW will be maintained throughout the intervention. Pedometers will be worn by participant in blind-mode throughout the intervention, and removed during exercise training sessions. Participants will enter information about whether they wore their pedometer on the study website. Aerobic exercise group participants will be told to make no conscious alterations to their physical activity or dietary habits
- Aerobic Exercise+ Physical Activity (AERO-PA): The goal of this group is to perform 6 months of aerobic exercise and increase the amount of physical activity outside of their training sessions. They will be asked to make no conscious changes to their dietary habits
  Aerobic Exercise+ Physical Activity: The Aerobic Exercise+ Physical Activity Group will participate in the same supervised exercise training intervention as the Aerobic Exercise Group, but will also increase the amount of non-exercise physical activity in their daily lives. After week 6 of intervention, participants will incrementally increase Non-Ex PA until they reach an average of 3,000 steps/day above baseline. Non-Ex PA will be increased with moderate physical activity consistent with daily living (i.e. leisurely walking in the evening, walking the dog etc.). Participants will also periodically have life-style counseling sessions with instructors with expertise in behavioral change support to their dietary habits
Period: Overall Study
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Started | 15 | 15 | 15
Completed | 14 | 12 | 13
Not Completed | 1 | 3 | 2
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Injury | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Aerobic Exercise Training | Aerobic Exercise+ Physical Activity | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 45
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (7.5) | 49.7 (6.5) | 54.1 (8.3) | 52.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 13 | 37
  Male | 4 | 2 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 7 | 4 | 14
  White | 12 | 8 | 11 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45
Weight [Mean (Standard Deviation); unit: kg] — Weight was measured on a scale at baseline and follow-up
  kg | 98.6 (12.8) | 102.9 (19.8) | 97.6 (8.6) | 99.7 (14.4)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 35.3 (3.8) | 36.6 (5.7) | 36.2 (5.0) | 36.0 (4.8)
Body fat percentage [Mean (Standard Deviation); unit: Percent] — Body fat was measured by dual x ray absorptiometry at baseline and follow-up. Body fat is expressed as percent of body mass that is fat compared to total mass
  Percent | 44.7 (4.7) | 46.1 (5.2) | 46.2 (6.0) | 45.7 (5.2)
Waist circumference [Mean (Standard Deviation); unit: cm] — Waist circumference was measured with a guilick tape measure. The distance around the waist was measured at the level of the umbilicus (belly button). This measurement was taken at baseline and follow-up
  cm | 106.8 (8.5) | 105.2 (10.5) | 103.6 (6.7) | 105.2 (8.6)
Absolute fitness [Mean (Standard Deviation); unit: L/min] — Absolute fitness describes the maximal amount of O2 consumed during a maximal exercise test. Fitness is measures by indirect calorimetry
  L/min | 2.0 (0.5) | 2.1 (0.6) | 2.0 (5.0) | 2.0 (5.0)
Relative Fitness [Mean (Standard Deviation); unit: mL/kg/min] — Relative fitness describes the the maximal amount of oxygen consumed during an maximal exercise test. This value is adjusted for the participants' body weight. This measurement is taken at baseline and follow-up
  mL/kg/min | 20.0 (4.6) | 20.3 (3.5) | 20.4 (3.0) | 20.2 (3.7)
Glucose [Mean (Standard Deviation); unit: mg/dL] — Describes blood glucose concentration from a blood sample. This measurement is taken at baseline and follow-up
  mg/dL | 96.4 (4.5) | 97.0 (6.8) | 96.3 (7.3) | 96.6 (6.2)
Insulin [Mean (Standard Deviation); unit: μU·mL-1] — Describes the concentration of insulin in the blood sample. This measurement is taken at baseline and follow-up
  μU·mL-1 | 17.1 (7.7) | 14.4 (5.8) | 17.1 (5.8) | 16.2 (6.5)
Very low density lipoprotein [Mean (Standard Deviation); unit: mg/dL] — Describes the concentration of very low density lipoprotein cholesterol in the blood. This is performed at baseline and follow-up
  mg/dL | 29.5 (12.8) | 23.6 (11.8) | 22.5 (9.7) | 25.2 (11.7)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Describes the concentration of cholesterol in the blood. This is performed at baseline and follow-up
  mg/dL | 189.0 (25.8) | 204.0 (25.5) | 208.1 (30.7) | 200.4 (28.1)
High density lipoprotein [Mean (Standard Deviation); unit: mg/dL] — Describes the concentration of high density lipoprotein cholesterol in the blood. This is performed at baseline and follow-up
  mg/dL | 47.3 (11.2) | 45.1 (8.8) | 58.1 (14.9) | 50.2 (12.9)
Low density lipoprotein [Mean (Standard Deviation); unit: mg/dL] — Describes the concentration of low density lipoprotein cholesterol in the blood. This is performed at baseline and follow-up
  mg/dL | 112.3 (23.9) | 204.0 (25.5) | 208.1 (30.4) | 200.4 (28.1)
Insulin Sensitivity [Mean (Standard Deviation); unit: index] — Insulin sensitivity was measured using an oral glucose tolerance test. With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Matsuda index. Insulin sensitivity was calculated with Matsuda index: [10,000 / √glucose minute 0 x insulin minute 0) (mean glucose (OGTT) x mean insulin OGTT)]. A higher result is better.
  index | 2.9 (1.4) | 4.9 (3.7) | 3.5 (1.5) | 3.7 (2.5)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Describes the concentration of triglycerides in the blood. This is performed at baseline and follow-up
  mg/dL | 147.7 (63.3) | 118.3 (59.1) | 112.9 (49.4) | 126.3 (58.4)
C-reactive protein [Mean (Standard Deviation); unit: mg/L] — measures the amount of c-reactive protein in the blood, which is a marker of inflammation. This was performed at baseline and follow-up
  mg/L | 1.8 (1.0) | 4.3 (3.5) | 4.0 (3.1) | 3.4 (3.0)
baseline steps [Mean (Standard Deviation); unit: steps/day] — The average of steps walked determined by accelerometry
  steps/day | 4479.3 (1285.9) | 4899.3 (1186.3) | 4528.3 (1296.0) | 4635.6 (1242.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Waist Circumference
Description: Waist circumference will be measured at the natural waist (midway between the inferior border of the rib cage and the superior aspect of the iliac crest) with a Gulick tape measure. Both landmarks (the inferior border of the ribcage and the superior aspect of the iliac crest) will be marked and the distance will be measured to determine the appropriate measurement site. Staff will confirm that: 1) the measurement tape remains horizontal; 2) the tape touches the entire circumference of the participant; 3) abdominal tissue is not compressed; 3) the tape measure is not within abdominal folds; 4) the measurement is taken at the end of normal respiration. The measurement will be repeated an additional time, and the reported value will be the average of these measurements. Both measurements must be within 0.5 cm to be considered acceptable for data purposes.
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | Control | Aerobic Exercise Training | Aerobic Exercise+ Physical Activity
Number analyzed (Participants) | 14 | 12 | 13
cm | -1.3 [-3.43 to 0.85] | -1.9 [-4.25 to 0.39] | -4.1 [-6.32 to -1.87]
Statistical Analysis 1: Comparison: Control vs Aerobic Exercise+ Physical Activity; Test type: Superiority; p = 0.074, ANCOVA
Statistical Analysis 2: Comparison: Control vs Aerobic Exercise Training; Change in waist circumference between AERO and CON; Test type: Superiority; p = 0.684, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training vs Aerobic Exercise+ Physical Activity; Comparison between the AERO group and the AERO-PA group; Test type: Superiority; p = 0.180, ANCOVA

2. Secondary Outcome: Change in Body Fat
Description: Dual-energy X-ray absorptiometry will be used to measure changes in fat and lean mass.
Time Frame: Baseline to 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of body fat
Arm/Group | Control | Aerobic Exercise Training | Aerobic Exercise+ Physical Activity
Number analyzed (Participants) | 14 | 12 | 13
percent of body fat | 0.071 [-0.68 to 0.82] | -0.71 [-1.53 to 0.09] | -1.35 [-2.13 to -0.57]
Statistical Analysis 1: Comparison: Control vs Aerobic Exercise+ Physical Activity; Change in body fat between the AERO-PA group and the CON group; Test type: Superiority; p = 0.011, ANCOVA
Statistical Analysis 2: Comparison: Control vs Aerobic Exercise Training; Test type: Superiority; p = 0.16, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training vs Aerobic Exercise+ Physical Activity; Change in body fat between the AERO and AERO-PA group; Test type: Superiority; p = 0.258, ANCOVA

3. Secondary Outcome: Change in Body Weight
Description: Weight will be measured using a standardized scale
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
kg | -0.44 [-2.01 to 1.20] | -1.11 [-2.88 to 0.66] | -2.38 [-4.08 to -0.68]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Comparison of body weight between the CON and AERO-PA groups; Test type: Superiority; p = 0.104, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in body weight between the CON and AERO groups; Test type: Superiority; p = 0.578, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in body weight between the AERO and AERO-PA groups; Test type: Superiority; p = 0.300, ANCOVA

4. Secondary Outcome: Change in Cardiorespiratory Fitness (L/Min)
Description: Fitness will be measured using a modified Balke protocol on a treadmill. Participants will walk at an initial speed of 2.0 mph with 0% grade for the first 3 minutes after which the treadmill speed will increase to 3.0 mph for the next 3 minutes. The treadmill grade will be increased by 2.5% every 3 minutes until volitional exhaustion. Respiratory gases (VO2, CO2) and ventilation will be measured continuously using a True Max 2400 Metabolic Measurement Cart (Parvomedics, Salt Lake City Utah).
Time Frame: Baseline and 24 weeks
Measure: Mean (95% Confidence Interval); unit: Liters/minute
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
Liters/minute | 0.01 [-0.11 to 0.12] | 0.094 [-0.04 to 0.22] | 0.28 [0.16 to 0.40]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in cardiorespiratory fitness (L/min) between the AERO and AERO-PA groups; Test type: Superiority; p = 0.002, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in cardiorespiratory fitness (L/min) AERO and CON groups; Test type: Superiority; p = 0.314, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in cardiorespiratory fitness (L/min) between the AERO and AERO-PA groups; Test type: Superiority; p = 0.041, ANCOVA

5. Secondary Outcome: Change in Insulin Sensitivity
Description: Insulin sensitivity was measured using an oral glucose tolerance test. With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Matsuda index. Insulin sensitivity was calculated with Matsuda index: [10,000 / √glucose minute 0 x insulin minute 0) (mean glucose (OGTT) x mean insulin OGTT)]. A higher result is better.
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Index
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
Index | 0.84 [-0.10 to 1.78] | 0.25 [-0.81 to 1.30] | 0.75 [-0.20 to 1.70]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in insulin sensitivity between the CON and AERO-PA groups; Test type: Superiority; p = 0.891, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in insulin sensitivity between the CON and AERO groups; Test type: Superiority; p = 0.417, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in insulin sensitivity between the AERO and AERO-PA groups; Test type: Superiority; p = 0.484, ANCOVA

6. Secondary Outcome: Change in Low Density Lipoprotein (LDL)
Description: LDL level will be measured from a blood sample at baseline and follow-up.
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
mg/dL | 2.2 [-11.6 to 16.0] | -5.2 [-20.1 to 9.6] | -8.7 [-22.9 to 5.6]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in Low density lipoprotein (LDL) between the CON and the AERO groups; Test type: Superiority; p = 0.274, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in Low density lipoprotein (LDL) between the CON and AERO groups; Test type: Superiority; p = 0.461, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in Low density lipoprotein (LDL) between AERO and AERO-PA groups; Test type: Superiority; p = 0.739, ANCOVA

7. Secondary Outcome: Change in High Density Lipoprotein (HDL)
Description: HDL cholesterol level will be measured from a blood sample at baseline and follow-up
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
mg/dL | -1.9 [-5.1 to 1.4] | -2.2 [-5.6 to 1.3] | -1.4 [-4.7 to 2.0]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in high density lipoprotein (HDL) between the CON and AERO-PA group; Test type: Superiority; p = 0.837, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in high density lipoprotein (HDL) between the CON and AERO groups; Test type: Superiority; p = 0.895, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Test type: Superiority; p = 0.744, ANCOVA

8. Secondary Outcome: Change in Total Cholesterol (mg/dL)
Description: Total cholesterol will be measured by a blood sample at baseline and 24 weeks
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
mg/dL | 6.1 [-7.6 to 19.9] | -5.4 [-20.3 to 9.4] | -12.3 [-26.6 to 1.9]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in total cholesterol (mg/dL); Test type: Superiority; p = 0.067, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in total cholesterol (mg/dL) between the CON and AERO groups; Test type: Superiority; p = 0.254, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in total cholesterol (mg/dL) between AERO and AERO-PA groups; Test type: Superiority; p = 0.501, ANCOVA

9. Secondary Outcome: Change in Triglyceride Level
Description: Change in triglycerides will be measured from a blood sample at baseline and 24 weeks
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
mg/dL | -1.6 [-20.6 to 17.5] | 9.6 [-10.9 to 30.2] | -11.7 [-31.5 to 8.0]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in triglyceride level between the AERO-PA and CON groups; Test type: Superiority; p = 0.456, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in triglyceride level between the CON and AERO groups; Test type: Superiority; p = 0.422, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in triglyceride level between the AERO and AERO-PA groups; Test type: Superiority; p = 0.136, ANCOVA

10. Secondary Outcome: Change in Glucose
Description: Glucose concentration from a fasting blood sample will be measured at baseline and follow-up
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
mg/dL | 1.0 [-2.2 to 4.2] | -1.6 [-5.1 to 1.9] | -0.62 [-3.9 to 2.7]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in glucose level between the CON and AERO-PA groups; Test type: Superiority; p = 0.483, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in glucose between the CON and AERO groups; Test type: Superiority; p = 0.274, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in glucose level between the AERO and AERO-PA groups; Test type: Superiority; p = 0.685, ANCOVA

11. Secondary Outcome: Change in C-reactive Protein
Description: High sensitivity c-reactive protein (inflammatory marker) will be measured at baseline and follow-up
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
mg/L | 0.83 [-0.16 to 1.83] | 0.51 [-0.57 to 1.58] | 0.34 [-0.69 to 1.37]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in systemic inflammation between CON and AERO-PA groups; Test type: Superiority; p = 0.489, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in systemic inflammation between the CON and AERO groups; Test type: Superiority; p = 0.652, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in systemic inflammation between the AERO and AERO-PA groups; Test type: Superiority; p = 0.822, ANCOVA

12. Secondary Outcome: Changes in Steps
Description: Participants will wear an accelerometer for seven consecutive days, 24-hrs/day. The amount of steps will be calculated
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
steps per day | -58.4 [-805.8 to 689.1] | 191.3 [-616.1 to 998.6] | 2324.5 [1548.9 to 3100.2]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Changes in steps between the CON group and the AERO-PA group; Test type: Superiority; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Changes in steps between the CON and the AERO group; Test type: Superiority; p = 0.648, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Changes in steps between the AERO and AERO-PA groups; Test type: Superiority; p < 0.001, ANCOVA

13. Secondary Outcome: Change in Caloric Intake (Kilocalories)
Description: Food Frequency Questionnaire (FFQ) contains approximately 105 items grouped by categories and is completed for both frequency of consumption as well as portion size selections by the individual. The questionnaire, upon completion, provides estimated daily intake values for selected nutrients (kilocalories, macronutrients, and micronutrients) and provides information on food group servings.
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: kcals
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
kcals | -553.2 [-874.7 to -231.6] | -264.3 [-599.0 to 70.3] | -276.9 [-589.4 to 44.6]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in kilocalories (dietary intake) between CON and AERO-PA group; Test type: Superiority; p = 0.226, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in caloric intake between the CON and the AERO groups; Test type: Superiority; p = 0.215, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in caloric intake (kilocalories) between the AERO and AERO-PA groups; Test type: Superiority; p = 0.957, ANCOVA

14. Secondary Outcome: Change in Insulin
Description: Insulin level will be measured from a fasting blood sample at baseline and at 24 weeks
Time Frame: Baseline and 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: μU·mL-1
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
Number analyzed (Participants) | 14 | 12 | 13
μU·mL-1 | -3.7 [-6.3 to -1.0] | -3.2 [-5.9 to -0.4] | -1.9 [-4.5 to 0.7]
Statistical Analysis 1: Comparison: Control (CON) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in insulin concentration between the CON and AERO-PA group; Test type: Superiority; p = 0.337, ANCOVA
Statistical Analysis 2: Comparison: Control (CON) vs Aerobic Exercise Training (AERO); Change in insulin level between the AERO and CON groups; Test type: Superiority; p = 0.770, ANCOVA
Statistical Analysis 3: Comparison: Aerobic Exercise Training (AERO) vs Aerobic Exercise+ Physical Activity (AERO-PA); Change in insulin concentration between AERO and AERO-PA groups; Test type: Superiority; p = 0.515, ANCOVA

ADVERSE EVENTS:
Time Frame: Data were collected over the course of approximately 6 month period that participants were enrolled. This included the assessment visits and the intervention
Arm/Group | Control (CON) | Aerobic Exercise Training (AERO) | Aerobic Exercise+ Physical Activity (AERO-PA)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-10-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT02010060/Prot_SAP_000.pdf
  • Informed Consent Form (2013-11-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT02010060/ICF_001.pdf